CLINICAL TRIAL: NCT00082147
Title: A Prospective Histopathologic Study of Dynamic Contrast Enhanced MRI for Prostate Cancer Delineation and Characterization With the APT-MRI System
Brief Title: Magnetic Resonance Imaging to Locate and Characterize Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 040171; 04-C-0171; NCT00085514 (obsolete NCT alias)
Record Dates: First submitted 2004-04-30; First posted 2004-04-30 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06-11

CONDITIONS: Prostate Cancer
Keywords: MRI; Biopsy; Fiducial Marker; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

ARMS (1):
- Biopsy (Experimental): Biopsy
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Patients will then undergo endorectal coil MR imaging of the prostate gland, including conventional anatomic imaging and dynamic-contrast-enhanced MRI During MR imaging, 4 to 10 needle biopsy cores of the prostate will be obtained using a trans-rectal needle guide system (APT-MRI).

SUMMARY:
This study will examine the usefulness of an imaging procedure called dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) for localizing and characterizing prostate cancer. For this test, a medicine is injected into a vein and the MRI measures how the medicine flows through the prostate gland. The measurements provide information about the blood vessels in the prostate gland, which provides other information about the cancer. Several needle biopsies are performed during the procedure, and the results of the biopsies are compared with the information from the DCE-MRI.

Men 18 years of age and older with suspected or confirmed prostate cancer may be eligible for this study. Candidates are screened with a medical history and physical examination, blood test, and review of tumor pathology.

Participants undergo DCE-MRI and needle biopsies of the prostate. The day before and the morning of the procedure, patients are given an antibiotic called Levofloxacin. They also have a small enema the morning of the test. A local anesthetic is then given in the area around the prostate to numb the tissue and decrease any discomfort from the procedure. A tube is placed in the rectum to obtain better pictures of the prostate gland during the imaging. During the scan, the patient may be asked to breathe air that contains higher concentrations of oxygen and carbon dioxide than are in room air. The MRI scans guide the physician in selecting areas of the prostate to biopsy. For each biopsy, a needle is placed through the rectum into the prostate gland. When the needle is in place, a small tissue sample is withdrawn. This procedure is repeated until 4 to 10 biopsies are taken. During the procedure, which lasts about 1 hour, the patient lies on his stomach on a stretcher.

Patients who are planning to undergo surgery or radiation treatment for their cancer at the NCI may have up to four 1-mm non-reactive gold markers placed in the prostate during the DCE-MRI procedure. The markers are left in place to help target the radiation treatments and to show where the biopsies were taken if the prostate is removed.

At the end of the procedure, the patient is moved to a bed to recover and may get up and urinate after about 30 to 60 minutes. After a period of observation, the patient is discharged home with a dose of antibiotic to take the next day.

Some patients may be asked to repeat the MRI and biopsy procedure during or after their treatment for prostate cancer to help investigators learn whether the MRI test is still helpful after treatment. Repeat testing is optional.

DETAILED DESCRIPTION:
Accurate spatial delineation and biologic characterization of tumors within the prostate gland by non-invasive means, such as MR imaging, stands to impact the spectrum of prostate cancer care. At present there are no imaging techniques that can accurately delineate tumor extent. With dynamic contrast enhanced MRI (DCE-MRI), signal intensity can be plotted over time for various regions of interest within the prostate, and reflect physiological parameters such as tissue perfusion, blood flow, vascular density and vascular permeability. Preliminary studies suggest that malignant tumors demonstrate a more rapid and intense uptake of contrast, as well as a more rapid washout compared with the normal peripheral zone. However, histopathologic confirmation of these findings has been limited.

This study strives to establish a correlation between K(trans) calculated from DCE-MRI data and the corresponding tissue histopathology. This will be achieved by acquiring needle biopsies with the APT-MRI (Access to Prostate Tissue under MRI-guidance) system in accurate spatial and temporal reference to DCE-MR images. The study will accrue 80 patients over a 2-year period with the primary analysis relating K(trans) to the probability of malignancy using Generalized Estimating Equations.

Patients who have undergone a TRUS-guided biopsy for suspected prostate cancer or patients with a pathological diagnosis of prostate cancer will be potential candidates for enrollment. Prior to the procedure, blood will be drawn and urine collected to measure PSA level and for protein profiling. Patients will then undergo endorectal coil MR imaging of the prostate gland, including conventional anatomic imaging and dynamic-contrast-enhanced MRI. During MR imaging, 4 to 10 needle biopsy cores of the prostate will be obtained using a trans-rectal needle guide system (APT-MRI). The ability to obtain prostate biopsy cores from all prostatic subzones and sites of interest will be documented, as will the overall procedure time and acute toxicities associated with the procedure. Histopathology and laboratory results of needle core biopsies will be compared to corresponding DCE-MRI measurements, prior TRUS-biopsy results, and/or prostatectomy specimens. This procedure may be repeated at a later time through the patient's course of observation, therapy, or follow up.

This is not a therapeutic trial. Patients admitted to this protocol will only be admitted to other protocols of experimental treatments if they also specifically meet the eligibility criteria for those protocols. Patients may derive benefit from the MRI-guided biopsy, which will be stated in the protocol consent document.

ELIGIBILITY:
* INCLUSION CRITERIA:
* ECOG performance status 0 or 1.
* Patients with a TRUS-guided biopsy for suspected prostate cancer in the past twelve months, or patients with pathologically confirmed adenocarcinoma of the prostate gland and who have not received definitive local therapy.
* Age greater than or equal to 18 years.
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

EXCLUSION CRITERIA:

* Contraindication to trans-rectal biopsy:
* Bleeding disorder;
* PT/PTT greater than or equal to 1.5 times the upper limit of normal;
* Platelets less than or equal to 50K;
* Active anticoagulation;
* Severe immunocompromise;
* Severe hemorrhoids;
* Surgically absent rectum.
* Contraindication to MRI:
* Patients weighing greater than 136 kgs (weight limit for the scanner tables);
* Allergy to MR contrast agent;
* Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI.
* Allergy to local anesthetics or quinolone antibiotics.
* Patients with a known diagnosis of prostate cancer and a known treatment plan to proceed to prostatectomy if the result of the biopsy would not affect surgical management.
* Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04-29; Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Correlation between the DCE-MRI kinetic parameter Ktrans and histopathologic determination of malignancy at corresponding biopsy sites within the prostate gland. | Post procedure

SECONDARY OUTCOMES:
To further determine the feasibility and tolerability of MRI-guided prostate biopsy with the APTMRI system. | completion of study
To determine the ability of the APT-MRI system to target all prostatic subzones and all sites suspicious of malignancy within the prostate gland. | completion of study
To obtain further data on the tissue targeting accuracy of the APT-MRI system for needle biopsy | completion of study
To determine if other DCE-MRI contrast kinetic parameters (Vf, amplitude, slope, and time to peak) correlate with the histopathologic determination of malignancy based on MRI-guided needle biopsies of the prostate gland. | completion of study
To determine if the subjective determination of malignant sites within the prostate gland based on DCE-MR images, T2W images, or both, correlates with the histopathologic determination of malignancy based on MRI-guided needle biopsies. | completion of study
To compare DCE-MRI data with the microvessel density of corresponding tissues. | completion of study
1.1.2.7 To compare DCE-MRI data with the microarray and proteomic profiles of corresponding tissues. | completion of study
To compare the histopathologic diagnosis and Gleason grade obtained with MRI-guided biopsies with prior TRUS-guided biopsy results. | completion of study
To compare the Gleason grade of MR-guided biopsies with the Gleason grade of prostatectomy specimens. | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Steineck G, Helgesen F, Adolfsson J, Dickman PW, Johansson JE, Norlen BJ, Holmberg L; Scandinavian Prostatic Cancer Group Study Number 4. Quality of life after radical prostatectomy or watchful waiting. N Engl J Med. 2002 Sep 12;347(11):790-6. doi: 10.1056/NEJMoa021483. PMID 12226149
- [Background] Potosky AL, Legler J, Albertsen PC, Stanford JL, Gilliland FD, Hamilton AS, Eley JW, Stephenson RA, Harlan LC. Health outcomes after prostatectomy or radiotherapy for prostate cancer: results from the Prostate Cancer Outcomes Study. J Natl Cancer Inst. 2000 Oct 4;92(19):1582-92. doi: 10.1093/jnci/92.19.1582. PMID 11018094
- [Background] Rabbani F, Stroumbakis N, Kava BR, Cookson MS, Fair WR. Incidence and clinical significance of false-negative sextant prostate biopsies. J Urol. 1998 Apr;159(4):1247-50. PMID 9507846